CLINICAL TRIAL: NCT00723203
Title: A Phase II Study of LBH589, a Novel Histone Deacetylase Inhibitor, in Relapsed and Refractory Adult Patients With Acute Leukemia (AL) or in Newly Diagnosed Patients Over the Age of 60
Brief Title: Panobinostat in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to a lack of efficacy
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07174; P30CA033572 (NIH); CHNMC-07174; NOVARTIS-CHNMC-07174; CDR0000601203 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Leukemia
Keywords: Philadelphia chromosome positive adult precursor acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Panobinostat; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (panobinostat) (Experimental): Patients receive oral panobinostat once on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  panobinostat: 40 mg Monday, Wednesday and Friday of every week in a 28 day cycle
  Interventions: Drug: panobinostat; Genetic: gene expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: panobinostat — 40 mg Monday, Wednesday and Friday of every week in a 28 day cycle
Genetic: gene expression analysis — Day 1 and day 28 samples
Genetic: reverse transcriptase-polymerase chain reaction — Day 1 and day 28 samples
Other: laboratory biomarker analysis — Day 1 and day 28 samples

SUMMARY:
RATIONALE: Panobinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying the side effects of panobinostat and to see how well it works in treating patients with relapsed or refractory acute lymphoblastic leukemia or acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the antitumor activity of panobinostat, in terms of objective response rate, time to progression, and survival, in patients with relapsed or refractory acute lymphoblastic leukemia or acute myeloid leukemia.
* To assess the toxicity of panobinostat in these patients.

Secondary

* To perform correlative laboratory studies to assess changes in various proteins that may be altered by histone deacetylase inhibition therapy.

OUTLINE: Patients receive oral panobinostat once on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo peripheral blood and bone marrow sample collection at baseline and on day 28 of course 1 for correlative laboratory studies. Samples are analyzed by RT-PCR for reactivation of FANCG, FOXO3A, GADD45A, GADD45B, GADD45G, H2AX, and TP73.

After completion of study treatment, patients are followed for at least 4 weeks.

PROJECTED ACCRUAL: A total of 74 patients (37 with acute myeloid leukemia and 37 with acute lymphoblastic leukemia) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed acute myeloid leukemia or acute lymphoblastic leukemia (ALL)

  * Relapsed or refractory disease
* Patients with Philadelphia chromosome-positive (Ph+) ALL refractory to BCR/ABL inhibitors are eligible
* Patients who have relapsed after prior autologous or allogenic stem cell transplant are eligible
* No active CNS disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Serum albumin ≥ 3 g/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (5.0 times ULN if transaminase elevation is due to leukemic involvement)
* Bilirubin ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 50 mL/min
* Potassium ≥ lower limit of normal (LLN)
* Phosphorous ≥ LLN
* Serum total calcium (corrected for serum albumin) or serum ionized calcium ≥ LLN
* Magnesium ≥ LLN
* Thyroid stimulating hormone and free T4 normal (thyroid hormone replacement therapy allowed)
* LVEF ≥ LLN by MUGA or ECHO
* No impaired cardiac function, including any of the following:

  * QTc > 450 msec
  * Congenital long QT syndrome
  * History of sustained ventricular tachycardia
  * History of ventricular fibrillation or torsades de pointes
  * Bradycardia (i.e., heart rate < 50 beats per minute)

    * Pacemaker allowed provided heart rate ≥ 50 beats per minute
  * Myocardial infarction or unstable angina within the past 6 months
  * New York Heart Association class III-IV congestive heart failure
  * Right bundle branch block and left anterior hemiblock (bifascicular block)
* No uncontrolled hypertension
* No unresolved diarrhea > CTCAE grade 1
* No impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral panobinostat
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 3 months after completion of study treatment
* No other primary malignancy within the past 5 years, other than curatively treated carcinoma in situ of the cervix or basal cell or squamous cell carcinoma of the skin
* No HIV or hepatitis C positivity
* No other concurrent severe and/or uncontrolled medical condition
* No significant history of non-compliance to medical regimens or inability to give reliable informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy
* More than 4 weeks since prior valproic acid
* No other prior treatment with a histone deacetylase inhibitor
* No concurrent medication that may cause QTc prolongation or induce torsades de pointes
* No concurrent CYP3A4 inhibitors
* No concurrent grapefruit, grapefruit juice, or Seville (sour) oranges
* No concurrent radiotherapy
* No other concurrent anticancer therapy or investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Popplewell, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - South Pasadena Cancer Center, Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Panobinostat): Patients receive oral panobinostat once on days 1, 3, and 5. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  panobinostat: 40 mg Monday, Wednesday and Friday of every week in a 28 day cycle
  gene expression analysis: Day 1 and day 28 samples
  reverse transcriptase-polymerase chain reaction: Day 1 and day 28 samples
  laboratory biomarker analysis: Day 1 and day 28 samples
Period: Overall Study
Arm/Group | Treatment (Panobinostat)
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Panobinostat)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 57 [19 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Hematological Response Rate
Description: Morphologic CR: morphologic leukemia-free state with absolute neutrophil count > 1000/uL and platelet count ≥ 100,000/uL and independent of blood transfusions. Cytogenic CR: morphologic CR along with reversion to a normal karyotype by cytogenetic analysis. Molecular CR: morphologic CR with no residual disease by molecular or flow cytometric detection methods. Morphologic CR with incomplete blood recovery (CRi): morphologic CR except for residual neutropenia (<1000/uL) and/or thrombocytopenia (<1000,000/uL). PR: same hematologic values for a CR but with a decrease of at least 50% in percentage of blasts to a post-treatment value of 5% to 25% in bone marrow aspirate. (If the pre-treatment blast percentage was 50-100% this must decrease to a value between 5-25%. If the pre-treatment blast percentage was 20-49% this must decrease by at least half to a value > 5%.) A value ≤ 5% is also considered a PR if Auer rods are present. Hematological response = morphologic CR+PR.
Time Frame: Up to 6 cycles of treatment, up to 24 weeks.
Population: Three patients of the 16 accrued were not included in the analysis for response per protocol due to patient refusal for alternative treatment prior to completing the first cycle of treatment.
Measure: Number; unit: percentage of responding participants
Arm/Group | Treatment (Panobinostat)
Number analyzed (Participants) | 13
percentage of responding participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a time period of 1 year and 9 months.
Description: "Other" adverse events includes all grades and attributions to treatment that are not included in "Serious" adverse events.
Arm/Group | Treatment (Panobinostat)
Serious Adverse Events (participants affected / at risk) | 11/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panobinostat) (N=16)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (3)
Disease progression (General disorders) | 5 (5)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 2 (3)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panobinostat) (N=16)
Hemoglobin decreased (Blood and lymphatic system disorders) | 16 (34)
Arrhythmia (Cardiac disorders) | 4 (8)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (3)
Cardiac disorder (Cardiac disorders) | 2 (2)
Nodal arrhythmia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Premature ventricular contractions (Cardiac disorders) | 3 (5)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 11 (17)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 2 (2)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (9)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 10 (14)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (13)
Oral hemorrhage (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Chest pain (General disorders) | 5 (5)
Chills (General disorders) | 7 (8)
Edema limbs (General disorders) | 3 (4)
Fatigue (General disorders) | 15 (28)
Fever (General disorders) | 6 (9)
Injection site reaction (General disorders) | 2 (2)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Hypersensitivity (Immune system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (4)
Alanine aminotransferase increased (Investigations) | 7 (10)
Alkaline phosphatase increased (Investigations) | 10 (20)
Aspartate aminotransferase increased (Investigations) | 6 (7)
Bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 5 (9)
Electrocardiogram QTc interval prolonged (Investigations) | 3 (4)
Fibrinogen decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (4)
Laboratory test abnormal (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 9 (22)
Lymphocyte count decreased (Investigations) | 6 (15)
Neutrophil count decreased (Investigations) | 10 (23)
Platelet count decreased (Investigations) | 13 (36)
Serum cholesterol increased (Investigations) | 1 (3)
Weight loss (Investigations) | 4 (5)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (10)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 6 (10)
Blood glucose increased (Metabolism and nutrition disorders) | 11 (20)
Blood uric acid increased (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 14 (24)
Serum calcium decreased (Metabolism and nutrition disorders) | 10 (21)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1)
Serum magnesium decreased (Metabolism and nutrition disorders) | 7 (14)
Serum magnesium increased (Metabolism and nutrition disorders) | 3 (4)
Serum phosphate decreased (Metabolism and nutrition disorders) | 6 (9)
Serum potassium decreased (Metabolism and nutrition disorders) | 6 (15)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 10 (15)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 8 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7)
Headache (Nervous system disorders) | 5 (5)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 2 (2)
Trigeminal nerve disorder (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4)
Protein urine positive (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 3 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (7)

LIMITATIONS AND CAVEATS:
There were no responses observed in the first 12 evaluable patients accrued to the first stage of the two-stage Optimum design of Simon. As a result the study was terminated due to a lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes